CLINICAL TRIAL: NCT03907891
Title: A Randomized Controlled Trial to Reduce Hopelessness Through Enhanced Physical Activity in Adults With Ischemic Heart Disease
Brief Title: Reducing Hopelessness Through Improved Physical Activity in Adults With Heart Disease: With COVID-19 Considerations
Acronym: Heart Up!
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Principal Investigator, Susan L Dunn, PhD, RN, FAHA, FAAN, Professor, University of Illinois at Chicago
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2018-1485; R01NR017649 (NIH); 3R01NR017649-04S1 (NIH)
Record Dates: First submitted 2019-04-03; First posted 2019-04-09 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Ischemic Heart Disease; Hopelessness; Physical Activity; Motivation; Social Support; Covid19
MeSH Terms: conditions — Myocardial Ischemia; Motor Activity; COVID-19

STUDY DESIGN:
Intervention Model Description: A three group RCT will be used to test the effectiveness of a mHealth intervention (Heart Up!) versus attention control to promote increased physical activity and reduce state hopelessness. Patients will be randomized to one of three groups: 1) motivational social support (MSS) from a nurse, 2) MSS from a nurse with additional significant other support (SOS), or 3) attention control (AC). Data will be collected at baseline, and 2, 6, 9 and 12 months.
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: The data collectors are also masked in the clinical trial.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Motivational social support (MSS) from a nurse alone (Experimental): Participants will receive a 60-minute session of motivational interviewing via videoconference or telephone (at participant discretion) in their home from a trained nurse. The nurse will apply motivational interviewing techniques to explore the patient's thoughts about making a behavior change to attain adequate physical activity (PA). Patients will be encouraged to exercise based on instructions provided by the hospital staff. The patient's ability to take their radial pulse before and after PA will be assessed, and patients will be provided written instructions on the correct manner to take a radial pulse. Patients will receive daily motivational text messages from the nurse for 6 weeks. The texts will be sent via the REDCap automated system. The automated system confirms that texts were sent. The motivational interviewer nurse will confirm by phone that the patient receives her/his first text from the REDCap system.
  Interventions: Behavioral: Motivational social support from nurse
- MSS from nurse with additional significant other support (SOS) (Experimental): Participants will also receive a 60-minute session of motivational interviewing via videoconference or telephone (at participant discretion) in their home from a trained nurse and text messages from a nurse for 6 weeks, as described in arm 1. In addition, patients will receive daily text messages from their significant other for 6 weeks. Researchers developed the 42 significant other text messages. The motivational interviewing nurse will provide the text messages to the significant other in writing. The order of texts sent from the significant other will be randomized so that we can determine their effectiveness in general. The significant other will be asked to type and send the text message listed for each date to the patient. Study staff will confirm by phone that the patient received the first text from the significant other. Patients will be asked to track the number of text messages from the significant other that they read over the 6-week period using the log provided.
  Interventions: Behavioral: Motivational social support from nurse with additional support from significant other
- Attention control (AC) (Active Comparator): Participants in the AC group will receive a 60-minutes session with a nurse via videoconference or telephone (at participant discretion) viewing of American Heart Association educational videos and and documents regarding IHD. The nurse will additionally provide a written copy of the hospital physical activity instructions, will assess the patient's ability to take their pulse, and provide written instructions on the correct manner to take a radial pulse.
  Interventions: Behavioral: Attention control

INTERVENTIONS:
Behavioral: Motivational social support from nurse — A 60-minute motivational interviewing session with a nurse, followed by 6 weeks of daily motivational social support text messages.
  Arms: Motivational social support (MSS) from a nurse alone
Behavioral: Motivational social support from nurse with additional support from significant other — A 60-minute motivational interviewing session with a nurse, followed by 6 weeks of daily motivational social support text messages from both a nurse and the patient's self-identified significant other.
  Arms: MSS from nurse with additional significant other support (SOS)
Behavioral: Attention control — A 60-minute session with a nurse focused on American Heart Association educational videos and written information.
  Arms: Attention control (AC)

SUMMARY:
After a 30-year decline, heart disease is projected to increase up to 18% by 2030. Participation rates in cardiac rehabilitation remain extremely low and hopeless individuals are less likely to participate. This innovative study has the potential to advance science, improve patient care, and improve patient outcomes by demonstrating the effectiveness of the Heart Up! program to increase physical activity and reduce hopelessness in patients with heart disease. Hopelessness is associated with a 3.4 times increased risk of mortality or nonfatal myocardial infarction in patients with ischemic heart disease (IHD), independent of depression. Hopelessness has been identified in 27-52% of patients with IHD and can persist for up to 12 months after hospital discharge. Hopelessness, a negative outlook and sense of helplessness toward the future, can be a temporary response to an event (state) or a habitual outlook (trait). Hopelessness is associated with decreased physical functioning and lower physical activity (PA) levels in individuals with IHD. While research has investigated strategies to increase PA among IHD patients in general, the study team is the only group to design an intervention to promote PA specifically in hopeless IHD patients. The purpose of this randomized controlled trial is to establish the effectiveness of our 6-week mHealth intervention (Heart Up!) to promote increased PA in hopeless patients with IHD. A total of 225 hopeless IHD patients will be enrolled from a large community teaching hospital in the Midwest. Patients will be randomized (75 per group) to one of three groups: 1) motivational social support (MSS) from a nurse, 2) MSS from a nurse with additional significant other support (SOS), or 3) attention control (AC). It is hypothesized that 1) The MSS with SOS group will have the greatest increase in average minutes of moderate to vigorous PA per day at 8 and 24 weeks as compared to the MSS only or AC groups; 2) Greater increase in minutes of moderate to vigorous PA per day will be associated with decreased state hopelessness levels from baseline to weeks 8 and 24; and 3) Increased social support and increased motivation will mediate the effects of Heart Up! on a greater increase in moderate to vigorous PA at 8 and 24 weeks. The findings from this study could transform care for IHD patients who are hopeless by promoting self-management of important PA goals that can contribute to better health outcomes.

DETAILED DESCRIPTION:
Hopelessness is associated with a 3.4 times increased risk of mortality or nonfatal myocardial infarction in patients with ischemic heart disease (IHD), independent of depression. Hopelessness has been identified in 27-52% of patients with IHD and can persist for up to 12 months after hospital discharge. Hopelessness, a negative outlook and sense of helplessness toward the future, can be a temporary response to an event (state) or a habitual outlook (trait). Hopelessness is associated with decreased physical functioning and lower physical activity (PA) levels in individuals with IHD. Low levels of PA independently contribute to increased death and adverse events in patients with IHD. Rates of PA in IHD patients continue to be unacceptably low in both hospital-based cardiac rehabilitation and home settings. Hopelessness frequently compounds this issue. The links among hopelessness, PA, and mortality and morbidity for patients with IHD remain unknown. While research has investigated strategies to increase PA among IHD patients in general, the study team is the only group to design an intervention to promote PA specifically in hopeless IHD patients. This research, based on Self Determination Theory and Cohen's Stress and Coping Social Support Theory, has shown feasibility and preliminary efficacy for a motivational intervention that integrates social support from both the patient's nurse and significant other to promote increased PA. The purpose of this randomized controlled trial is to establish the effectiveness of our 6-week mHealth intervention (Heart Up!) to promote increased PA in hopeless patients with IHD. The study team will enroll 225 hopeless IHD patients from a large community teaching hospital in the Midwest. Patients will be randomized (75 per group) to one of three groups: 1) motivational social support (MSS) from a nurse, 2) MSS from a nurse with additional significant other support (SOS), or 3) attention control (AC). Data will be collected at baseline, months 2, 6, 9 and 12 using an accelerometer for PA and valid and reliable instruments of physical and emotional health and behaviors. The specific aims are to: 1) test the effectiveness of 6 weeks of MSS and MSS with SOS on increasing mean minutes per day of moderate to vigorous PA, measured by an ActiGraph accelerometer; 2) determine the effects of change in minutes per day of moderate to vigorous PA on state hopelessness, measured by the State-Trait Hopelessness Scale; and 3): determine if social support (measured by the ENRICHD Social Support Inventory) and motivation (measured by the Exercise Self-Regulation Questionnaire) mediate the effects of the Heart Up! intervention on PA. The specific aims of the supplement are to: 1) determine how the potentially negative impact of COVID-19 shelter-in-place/physical distancing measures on mental, social, and behavioral health outcomes are limited (moderated) by the RCT intervention and 2) using the Coronavirus Impact Scale, we will determine how the direct impact of COVID-19 life changes on mental, social, and behavioral health outcomes are limited (moderated) by the RCT intervention. The findings from this study could transform care for IHD patients who are hopeless by promoting self-management of important PA goals that can contribute to better health outcomes. This proposal supports NINR's investment in self-management to improve the quality of life for individuals with chronic illness.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥18 years old
* Diagnosed with MI, unstable angina, who undergo percutaneous coronary intervention (PCI) or coronary artery bypass graft (CABG) surgery
* Use a cell phone with text messaging
* Receive a recommendation to engage in physical activity either at home or in a hospital-based cardiac rehabilitation setting
* Have a planned discharge home
* Can identify a significant other who can text message them
* Speak and read English
* Can complete the screening instrument
* A score of ≥1.8 on the 10-item state subscale of the State-Trait Hopelessness Scale

Exclusion Criteria:

• None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 225 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2024-09-16 (Actual); Study Completion 2024-09-16 (Actual)

PRIMARY OUTCOMES:
ActiGraph GT9X Link Accelerometer | Month 12
  Mean minutes/day moderate to vigorous physical activity
State-Trait Hopelessness Scale | Month 12
  Participant's report of current level of state hopelessness. Total score range= 1 (better) to 4 (worse).

SECONDARY OUTCOMES:
Exercise Self-Regulation Questionnaire | Month 12
  Participant's report of exercise self-regulation level. Total score range= 1 (worse) to 7 (better).
ENRICHD Social Support Inventory | Month 12
  Participant's report of perceived social support level. Total score range= 1 (worse) to 30 (better).

OTHER OUTCOMES:
Charlson Comorbidity Index | Week 1
  Comorbidity score based on medical record abstraction. Total score range= 0 (better) to 100 (worse).
Cardiac Rehabilitation Exercise Participation Tool | Month 12
  Participant's report of participation level with exercise in home, community or cardiac rehabilitation program
Patient Health Questionnaire-9 | Month 12
  Participant's report of mean level of depressive symptoms. Total score range= 0 (better) to 27 (worse).
PROMIS-29 | Month 12
  Participant's report of mean level of well-being. Total score range= 4 (better) to 20 (worse).
Snyder State Trait Scales | Month 12
  Participant's report of mean level state and trait hope. Total score range= 8 (worse) to 64 (better).
EuroQol (EQ-5d-5L) | Month 12
  Participant's report of mean level of quality of life. Total score range= 1 (better) to 5 (worse).
Multi-Ethnic Study of Atherosclerosis (MESA) COVID-19 Questionnaire | Month 12
  Participant's report of COVID-19 symptoms, diagnosis, testing, and social distancing. No score range (14 items).
Coronavirus Impact Scale | Month 12
  Participant's report of impact on routine; income/ employment; access to food, medical and mental health care, extended family; and stress. No range (12 items)

CONTACTS AND LOCATIONS:
Overall Officials: Susan L Dunn, PhD, Principal Investigator — University of Illinois at Chicago
Locations (1):
- Spectrum Health, Grand Rapids, Michigan, United States

IPD SHARING:
Plan to Share IPD: Yes
Researchers will adhere to the NIH Policy on the Dissemination of NIH-Funded Clinical Trial Information. Data sets and associated documentation will be provided. The data sets will include data from questionnaires, the motivational intervention, and accelerometer-measured physical activity raw data elements and summary information. The dataset will be prepared in accordance with guidelines for the data repository. Key study documents (e.g., protocols, procedures, and instruments) that will enable the use of prepared data sets by outside investigators will be provided. A summary documentation file will be created to provide a complete overview of the data and a description of their use for investigators who are not familiar with the data set.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Summary results information from the clinical trial will be submitted to ClinicalTrials.gov no later than 12 months after the trial's completion date.
Access Criteria: Data will only be made available under terms and conditions consistent with the informed consent provided by the individual participants, and as approved by the UIC IRB and any local, state, and federal laws and regulations. Requests can be made directly to the PI, who will review requests.

REFERENCES:
- [Background] Dunn SL, DeVon HA, Collins EG, Luong A, Buursma MP, Gutierrez-Kapheim M, Bronas UG. Suicide Risk Management Protocol for a Randomized Controlled Trial of Cardiac Patients Reporting Hopelessness. Nurs Res. 2021 Jan/Feb;70(1):72-79. doi: 10.1097/NNR.0000000000000474. PMID 32956255
- [Background] Dunn SL, Robbins LB, Tintle NL, Collins EG, Bronas UG, Goodyke MP, Luong A, Gutierrez-Kapheim M, DeVon HA. Heart up! RCT protocol to increase physical activity in cardiac patients who report hopelessness: Amended for the COVID-19 pandemic. Res Nurs Health. 2021 Apr;44(2):279-294. doi: 10.1002/nur.22106. Epub 2021 Jan 11. PMID 33428224
- [Background] Luong A, Goodyke M, Dunn SL, Baynard T, Bronas U. ActiGraph and Short-term Heart Rate Variability Study Protocol: Amended for the COVID-19 Pandemic. J Cardiovasc Nurs. 2021 Nov-Dec 01;36(6):599-608. doi: 10.1097/JCN.0000000000000817. PMID 33833190
- [Derived] Goodyke MP, Tintle N, Collins E, DeVon HA, Bronas UG, Baynard T, Dunn SL. Lower Perceived Social Support Associated With Greater Hopelessness in Patients After an Acute Ischemic Heart Disease Event. J Cardiovasc Nurs. 2025 Sep-Oct 01;40(5):E239-E247. doi: 10.1097/JCN.0000000000001163. Epub 2024 Oct 24. PMID 39454079
- [Derived] Goodyke MP, Bronas UG, Baynard T, Tintle N, DeVon HA, Collins E, Dunn SL. Relationships Among Heart Rate Variability, Perceived Social Support, and Hopelessness in Adults With Ischemic Heart Disease. J Am Heart Assoc. 2024 Feb 20;13(4):e032759. doi: 10.1161/JAHA.123.032759. Epub 2024 Feb 13. PMID 38348815